CLINICAL TRIAL: NCT03764709
Title: The Technological Challenge of Continuous Wireless Monitoring in Internal Medicine Unit to Improve Management of Complex Patients: the Green Line From Hospital to Territory (Green Line H-T Study)
Brief Title: Continuous Wireless Monitoring in Internal Medicine Unit: the Green Line From Hospital to Territory
Acronym: GreenLightHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale del Garda (Other Government)
Collaborators: ASL Roma 6 (Other)
Responsible Party: Principal Investigator, Filomena Pietrantonio, Internal Medicina unit Director, Azienda Socio Sanitaria Territoriale del Garda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Green Light HT 2018
Record Dates: First submitted 2018-08-28; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Patient Monitoring
Keywords: Wireless monitoring, hospital-territory integration

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open-label, monocentric study for the evaluation of two different settings of critically ill patients recovered in Internal Medicine unit (IMU) and subsequently sent to subacute managed care unit or to earlier discharge, in order to evaluate the effectiveness of a wireless monitoring of clinical conditions vs. a traditional clinical monitoring on outcomes (critical adverse events, clinical exacerbations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vital signs wireless monitoring system GROUP A (Experimental): GROUP A clinical hypothesis: reduction in the number of exacerbations in stable inpatients who transit towards subacute managed care unit.
  The experimental arm will wear wireless monitoring for 5 days after transfer in subacute care unit
  Interventions: Device: Vital signs wireless monitoring system
- Control arm GROUP A (Active Comparator): GROUP A clinical hypothesis: reduction in the number of exacerbations in stable inpatients who transit towards subacute managed care unit.
  The active comparator arm will be monitored by nursing staff.
  Interventions: Device: Vital signs wireless monitoring system
- Vital signs wireless monitoring system GROUP B (Experimental): GROUP B clinical hypothesis: non-inferiority in the number of major clinical complications that, if treated at an earlier stage, can improve outcomes in stable patients who are selected for earlier discharge and are followed by a remote wireless monitoring at home.
  The experimental arm will wear wireless monitoring for 5 days after discharge at home
  Interventions: Device: Vital signs wireless monitoring system
- Control Arm GROUP B (Active Comparator): GROUP B clinical hypothesis: non-inferiority in the number of major clinical complications that, if treated at an earlier stage, can improve outcomes in stable patients who are selected for earlier discharge and are followed by a remote wireless monitoring at home.
  The active comparator arm will perform usual checks by caregivers at home.
  Interventions: Device: Vital signs wireless monitoring system

INTERVENTIONS:
Device: Vital signs wireless monitoring system — WIN@Hospital wireless remote monitoring is a modern light monitoring medical device with no need for continuous presence of a dedicated person. WIN@Hospital is based on an innovative modular and wearable device laid out for remote monitoring of several vital parameters 24/7. Dexcom G6 is a continuous glucose monitoring system which measures interstitial fluid glucose levels in people with diabetes from a sensor applied to the skin as an alternative to routine finger-prick blood glucose testing, and can produce a -continuous record of measurements which can be checked using an App. It can also indicate glucose level trends over time. Monitoring devices will be applied to all patients randomly assigned to the wireless monitoring arm, with a continuous monitoring setting over the first 5 days after the initiation of monitoring, corresponding to the starting of the observation (i.e. transition to subacute unit for GROUP A, discharge for GROUP B).

SUMMARY:
Study Information Indication* This is a prospective, randomized, controlled, open-label, monocentric study for the evaluation of two different settings of critically ill patients recovered in Internal Medicine unit (IMU) and subsequently sent to subacute managed care unit or to earlier discharge, in order to evaluate the effectiveness of a wireless monitoring of clinical conditions vs. a traditional clinical monitoring on outcomes (critical adverse events, clinical exacerbations).

Phase*: 4, observational prospective

Number of subjects*:

GROUP A and GROUP B: N=300 patients (150 per arm)

DETAILED DESCRIPTION:
Background and Rationale* In IMU there is an increasing concentration of patients with serious illness, under acute exacerbation of previous diseases, elderly patients with co-morbidities and/or fragility, needing high intensity care. Those patients need an overall evaluation of the rank of severity, complexity and dependence of their pathology, together with an evaluation of their risk of clinical deterioration, to implement a stratification of optimal treatments, intensity of care, length of stay. This could allow to optimize the approach to the complexity of the patients while helping containing costs, not only on the patients who are evaluated during their stay in IMUs, but also in those patients who undergo protected hospital discharge or transition to subacute intensive care unit.

Objectives*

Some preliminary data on wireless monitoring in IMU have shown that the timely identification of clinical instability could led to a shorter length of stay. Monitoring on clinically unstable patients lets to prevent the deterioration of adverse events, thus allowing a rapid onset of intervention. There are some expected outcomes following the adoption of a wireless clinical monitoring system:

1. Shorter length of stay and earlier discharge
2. Lower transition rate to Intensive Care Unit (ICU)
3. Earlier transition of patients from higher to lower intensity of care
4. Shorter time needed by nurses for the detection of vital signs and clinical parameters, and possibility to dedicate to high-quality activities

Therefore the present study aims to provide data regarding the impact of a specific and oriented integrated remote system for the monitoring of vital status of critically ill patients in the improvement of outcomes and in a more efficient prevision of length of stay and costs, and to verify whether the regular use of a wireless remote monitoring system could improve the quality of the assistance and reduce major complications vs. a traditional monitoring of clinical status executed by the nursing staff, in two specific settings of critically ill patients referring to Internal Medicine with acute conditions:

GROUP A: Patients who undergo a transition to a subacute intensive care unit, in terms of reduction of re-exacerbation, re-access to emergency department or need of intervention by Internal Medicine unit specialists by the use of wireless monitoring vs. traditional monitoring.

GROUP B: Patients who are selected for an earlier discharge from Internal Medicine Unit, in terms of non-inferiority in the incidence of major clinical complications.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients admitted to the Internal Medicine Unit regardless of the reason for admission.

  2. For GROUP A: eligibility to the transition towards subacute managed care unit (based on clinical evaluation).

  3. For GROUP B: eligibility to early discharge based on clinical evaluation and stable MEWS/NEWS scores.

Exclusion Criteria:

* - Inability to discernment
* Lack of informed consent/unwillingness to participate
* MEWS/NEWS out of range
* Transition to rehabilitation, Hospice, RSA or other Acute unit
* Pacemaker carriers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-27 (Estimated); Primary Completion 2021-01-27 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Major complications' reduction | 24 months
  Difference in the incidence of major complications 30 days after the transfer from the acute to the subacute areas and from the hospital to home among the patients subjected to continuous telemonitoring and those subjected to standard monitoring.

SECONDARY OUTCOMES:
% of early discharge | 24 months
  Percentage of patients admitted to acute medicine who reach the 7-day transfer criteria in the ward for subacutes and percentage of patients admitted to acute medicine who reach the criteria for discharge at home within 7 days
% of late major complications | 24 months
  3. Difference in the incidence of major complications at the conclusion of the standard telemonitoring / clinical monitoring phase 30 after the transfer from the acute to the subacute UOC and from the hospital to the home among the patients subjected to continuous telemonitoring and those subjected to standard monitoring .
Complications' risk factors | 24 months
  Patients'characteristics who predispose to major complications

CONTACTS AND LOCATIONS:
Locations (1):
- ASL Roma6, Albano Laziale, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] F. Pietrantonio, L. Piasini, F. Spandonaro. Internal Medicine and emergency admissions: from a national Hospital Discharge Records (SDO) study to a regional analysis. Italian Journal of Medicine Italian Journal of Medicine 2016; volume 10:157-167
- [Background] Blais R, Sears NA, Doran D, Baker GR, Macdonald M, Mitchell L, Thales S. Assessing adverse events among home care clients in three Canadian provinces using chart review. BMJ Qual Saf. 2013 Dec;22(12):989-97. doi: 10.1136/bmjqs-2013-002039. Epub 2013 Jul 4. PMID 23828878
- [Background] Sears N, Baker GR, Barnsley J, Shortt S. The incidence of adverse events among home care patients. Int J Qual Health Care. 2013 Feb;25(1):16-28. doi: 10.1093/intqhc/mzs075. Epub 2013 Jan 2. PMID 23283731
- [Background] Pietrantonio F, Orlandini F, Moriconi L, La Regina M. Acute Complex Care Model: An organizational approach for the medical care of hospitalized acute complex patients. Eur J Intern Med. 2015 Dec;26(10):759-65. doi: 10.1016/j.ejim.2015.08.011. Epub 2015 Sep 11. PMID 26365373
- [Background] Masotti P, McColl MA, Green M. Adverse events experienced by homecare patients: a scoping review of the literature. Int J Qual Health Care. 2010 Apr;22(2):115-25. doi: 10.1093/intqhc/mzq003. Epub 2010 Feb 10. PMID 20147333
- [Background] Doran D, Hirdes JP, Blais R, Baker GR, Poss JW, Li X, Dill D, Gruneir A, Heckman G, Lacroix H, Mitchell L, O'Beirne M, Foebel A, White N, Qian G, Nahm SM, Yim O, Droppo L, McIsaac C. Adverse events associated with hospitalization or detected through the RAI-HC assessment among Canadian home care clients. Healthc Policy. 2013 Aug;9(1):76-88. PMID 23968676
- [Background] Vincent C, Amalberti R. Safer Healthcare: Strategies for the Real World [Internet]. Cham (CH): Springer; 2016. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK481869/ PMID 29465922
- [Background] F. Pietrantonio. Analisi dei modelli esistenti: Acute Complex Care Model (ACCM). QUADERNI - Italian Journal of Medicine 2018; volume 6(3):18-29
- [Background] Brown H, Terrence J, Vasquez P, Bates DW, Zimlichman E. Continuous monitoring in an inpatient medical-surgical unit: a controlled clinical trial. Am J Med. 2014 Mar;127(3):226-32. doi: 10.1016/j.amjmed.2013.12.004. Epub 2013 Dec 14. PMID 24342543
- [Background] Tartaglia R, Albolino S, Bellandi T, Bianchini E, Biggeri A, Fabbro G, Bevilacqua L, Dell'erba A, Privitera G, Sommella L. [Adverse events and preventable consequences: retrospective study in five large Italian hospitals]. Epidemiol Prev. 2012 May-Aug;36(3-4):151-61. Italian. PMID 22828228
- [Background] Charles V. Sicurezza del paziente. Edizione italiana a cura di Tartaglia R, Albolino S, Bellandi T. Milano, Springer-Verlag Italia, 2012
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Background] Bellocco A. Risk management in ospedale. Risk News CINEAS (Consorzio Universitario per l'Ingegneria nelle Assicurazioni) 2002;23.
- [Background] Sensium Science MF06-01, April 2015
- [Background] Miglioramento della qualità della vita dei pazienti e riduzione del costo per il SSN attraverso l'uso di un sistema wireless di monitoraggio multi-parametrico dei parametri fisiologici. Case study sull'adozione del sistema di monitoraggio fisiologico WIN@Hospital presso l'Ospedale Campo di Marte, Lucca. Cangemi A, Turchetti B. Europe Health Summit Berlino (4-8 Maggio 2014)